CLINICAL TRIAL: NCT01437020
Title: A Phase I/II Clinical Trial To Assess the Safety and Biologic Activity of the Anti-IL-10 Monoclonal Antibody, SCH708980, in Combination With AmBisome(Registered Trademark), Versus That of Placebo in Combination With Ambisome(Registered Trademark), in Subjects With Visceral Leishmaniasis (VL)
Brief Title: SCH708980 With and Without AmBisome for Visceral Leishmaniasis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Drug Product no longer available.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-I-N222; 11-I-N222 (Other: NIH)
Record Dates: First submitted 2011-09-16; First posted 2011-09-20 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Leishmaniasis; Effects of Immunotherapy
Keywords: IL-10; Leishmaniasis; Immunotherapy
MeSH Terms: conditions — Leishmaniasis | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose escalating-IV infusion of SCH708980 and Ambisome (Experimental)
  Interventions: Drug: SCH708980 Anti-IL-10 monoclonal; Drug: AmBisome

INTERVENTIONS:
Drug: SCH708980 Anti-IL-10 monoclonal — Participants in Part 1 of the study will receive varying doses (0.3 mg/kg, 1.0 mg/kg, 3.0 mg/kg, or 10.0 mg/kg) of a single IV infusion of SCH708980. Participants in Part 2 of the study will receive a single IV infusion of SCH708980 on Day 1.
Drug: AmBisome — Participants in Part 1 of the study will receive a single IV infusion of AmBisome (10 mg/kg) 7 days after they receive SCH708980. Participants in Part 2 of the study will receive varying doses (3.75 mg/kg, 5 mg/kg, or 10 mg/kg) of a single IV infusion of AmBisome on Day 8.

SUMMARY:
Background:

- Visceral leishmaniasis (VL) is an infection caused by parasites carried by sand flies. The parasites cause fever, weight loss, and enlargement of the spleen and liver. They can also affect the blood and immune system. One possible treatment for VL involves an experimental drug called SCH708980, which may help to prevent the immune system from becoming suppressed and worsening the VL. Researchers want to give the drug along with AmBisome(Registered Trademark), which kills the parasites, to see if it is a safe and effective treatment.

Objectives:

- To study the safety and effectiveness of SCH708980, alone and combined with AmBisome(Registered Trademark), as a treatment for visceral leishmaniasis.

Eligibility:

* Individuals 18 to 60 years of who have been diagnosed with visceral leishmaniasis in the past 4 to 5 days, are HIV-negative, and are willing to stay in the hospital for 30 days.
* All participants will come from and be treated at the Kala-Azar Medical Research Center in Muzaffarpur, India.

Design:

* This is a two-part study. Participants will be assigned to only one part of the study.
* Participants will be screened with a medical history and physical exam; blood, urine, and stool samples, spleen or bone marrow samples; spleen measurements; a chest xray; and a heart function test.
* Part 1 participants will be separated into two groups: a larger group will have a selected dose of the study drug followed by AmBisome 7 days later, and a smaller group will have a placebo treatment followed by AmBisome.
* Part 2 participants will have either the study drug or a placebo plus AmBisome, based on the test results from the Part 1 participants.
* All participants will be monitored in the hospital for 30 days, and will have the following tests:
* Regular blood samples
* Urine and stool samples (day 14)
* Spleen measurements (days 8, 14, 21, and 30)
* Spleen or bone marrow sample (day 30 only). Participants who still have VL symptoms will give another sample on day 45.
* At 6 months after the start of treatment, participants will have a follow-up visit with spleen measurements, blood and stool samples, and possible spleen or bone marrow samples

DETAILED DESCRIPTION:
Visceral leishmaniasis (VL) or kala-azar is the most severe form of leishmaniasis, which can be fatal if left untreated. The majority of VL cases are found in resource-poor regions, including India (Bihar), Bangladesh, Brazil, Nepal, and Sudan. VL pathogenesis has been linked to an overproduction of the anti-inflammatory cytokine, interleukin (IL)-10, which can promote parasite replication and disease progression. Experimental models have shown that IL-10 plays a key role in the pathogenesis of VL.

The current study has two parts. Part 1 will be an open-label, dose-escalating design to determine the safety and tolerability of SCH708980 used in combination with AmBisome(Registered Trademark). Part 2 will be a randomized, single-blind, placebo-controlled, parallel design. A total of 50 subjects (n=10 subjects/group) will be enrolled in part 1 of the study. A group of 10 subjects will be observed for 7 days prior to receiving AmBisome(Registered Trademark) (10 mg/kg) on the 8th day, as part of the control group. Subsequently, 40 subjects (10 subjects/group) will receive a single intravenous (IV) infusion of SCH708980 (0.3 mg/kg, 1.0 mg/kg, 3.0 mg/kg, or 10 mg/kg) followed by a single IV infusion of AmBisome(Registered Trademark) (10 mg/kg) 7 days later. The first 2 subjects from each dose group to receive SCH708980 will be followed for 3 days after the drug is administered before treatment is initiated in the remaining 8 subjects in that group. Also, all individuals in each group will be followed for 7 days after AmBisome(Registered Trademark) is administered before the next higher dose-level group is enrolled in the study. Dose escalation will continue to the next dose level unless dose-limiting toxicities occur in > 20% of subjects in any cohort.

The dose level of SCH708980 to use in part 2 of the study will be decided 30 days after the start of AmBisome(Registered Trademark) treatment in the group receiving the highest dose in part 1. Randomization and accrual for part 2 of the study will begin at this time. The highest safe dose of SCH709890 (< 20% of subjects with dose-limiting toxicity) will be administered to subjects, not to exceed 10 mg/kg. Thirty subjects (n=10 subjects/group) will be randomized to 1:1:1 to receive:

1. A single IV infusion of SCH708980 (less than or equal to 10.0 mg/kg) on day 1 followed by a single IV infusion of AmBisome(Registered Trademark) (3.75 mg/kg) on day 8.
2. A single IV infusion of SCH708980 (less than or equal to 10.0 mg/kg) on day 1 followed by a single IV infusion of AmBisome(Registered Trademark) (5 mg/kg) on day 8.
3. A single dose of placebo on day 1 followed by a single IV infusion of AmBisome(Registered Trademark) (10 mg/kg) on day 8.

SCH709890 and placebo will be administered over 60 minutes, while AmBisome(Registered Trademark) will be administered over 120 minutes.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects (18 to 60 years of age) who meet the following criteria are eligible to enter the study:

* Newly diagnosed VL (within 4 to 5 days of screening) and confirmed by spleen or bone marrow aspirate.
* Clinical signs and symptoms compatible with VL: fever (> 99 degrees F) over a 2-week duration, splenomegaly (palpable spleen below the costal margin), and weight loss.
* Biochemical and hematological test values:

Hemoglobin > 6.0g/100mL.

WBC count > 1.0 times 10(9)/L.

Platelet count > 40 times 10(9)/L.

Aspartate aminotransferase (AST),alanine transaminase (ALT), and alkaline phosphatase < 3 times the upper limit of normal.

Prothrombin time (PT) < 4 seconds above the control values.

Serum creatinine levels within normal limits (males, 0.7 mg/dL - 1.1 mg/dL; females, 0.6 mg/dL - 0.9 mg/dL).

* Human immunodeficiency virus (HIV)-negative status.
* Willingness to be hospitalized for 30 days.
* Willingness to have samples stored.
* Negative serum pregnancy test result for women of childbearing potential.

EXCLUSION CRITERIA:

* A history of intercurrent or concurrent diseases (e.g., chronic alcohol consumption or drug addiction; renal, hepatic, cardiovascular, or central nervous system disease; diabetes; tuberculosis or other infectious or major psychiatric diseases) that may introduce variables affecting the outcome of the study.
* Any condition which, in the investigator's opinion, may prevent the subject from completing the study and the subsequent follow-up.
* Previous treatment for VL within 45 days of study enrollment.
* A history of allergy or hypersensitivity to amphotericin B.
* Prior treatment failures with amphotericin B.
* Current use of other drugs with known anti-leishmanial activity (e.g., antimonials, pentamidine, paromomycin, miltefosine), azoles (e.g., fluconazole, ketoconazole or itraconazole), nephrotoxic drugs, immunosuppressive drugs, other investigational agents, immunomodulatory drugs.
* Breastfeeding women
* Vaccinations within 30 days prior to enrollment in the study.

Exclusion of children:

Subjects younger than 18 years of age will be excluded from the study because insufficient data are available supporting dosing with SCH708980 in adults to judge the potential risk in children.

Exclusion of women:

Pregnant and lactating women are excluded from the study because insufficient data are available supporting dosing with SCH708980 in these populations to judge the potential risk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of a single IV infusion of SCH708980 (0.3 mg/kg, 1.0 mg/kg, 3 mg/kg, or 10 mg/kg) over the initial 7 days and in combination with a single IV infusion of AmBisome® (10 mg/kg) on the 8th day in part 1 of the study | Measured through Day 8

SECONDARY OUTCOMES:
The anti-IL-10 parasitic effect, as measured by real-time polymerase chain reaction (RT-PCR) | Measured 6 months after the start of treatment
Serum concentrations of SCH708980 | Measured 6 months after the start of treatment
Clinical response | Measured 6 months after the start of treatment
Outcomes at 6 months post-treatment | Measured 6 months after the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Sundar, MD, Principal Investigator — Institute of Medical Sciences, Banaras Hindu Universtiy, Varanasi, India; David Sacks, PhD, Principal Investigator — Laboratory of Parasitic Diseases, NIAID, NIH
Locations (2):
- India (2):
  - Kala-Azar Medical Research Center (KAMRC), Rambag Road, Muzaffarpur
  - Banaras Hindu University, Varanasi

REFERENCES:
- [Background] Desjeux P. Leishmaniasis. Public health aspects and control. Clin Dermatol. 1996 Sep-Oct;14(5):417-23. doi: 10.1016/0738-081x(96)00057-0. No abstract available. PMID 8889319
- [Background] Addy M, Nandy A. Ten years of kala-azar in west Bengal, Part I. Did post-kala-azar dermal leishmaniasis initiate the outbreak in 24-Parganas? Bull World Health Organ. 1992;70(3):341-6. PMID 1638662
- [Background] Bern C, Hightower AW, Chowdhury R, Ali M, Amann J, Wagatsuma Y, Haque R, Kurkjian K, Vaz LE, Begum M, Akter T, Cetre-Sossah CB, Ahluwalia IB, Dotson E, Secor WE, Breiman RF, Maguire JH. Risk factors for kala-azar in Bangladesh. Emerg Infect Dis. 2005 May;11(5):655-62. doi: 10.3201/eid1105.040718. PMID 15890115